CLINICAL TRIAL: NCT06291649
Title: Multicentre Prospective Observational Study of Acute Intoxications in Paediatric Age
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Marco De Luca, Principal Investigator, Meyer Children's Hospital IRCCS
Other Study IDs: AMIETOX
Record Dates: First submitted 2024-02-15; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Acute Intoxication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute intoxications represent a major public health problem, especially when affect a population such as children, who are vulnerable and at greater risk of unintentional and preventable poisonings.

The primary objective of the study is to assess the epidemiology of acute intoxications in paediatric age with respect to the social and care factors associated with it in order to then implement in the future a better diagnostic-therapeutic management modality on a national level.

Thi is a prospective non-profit multicentre observational cohort study on acute intoxications in the paediatric age, conducted by AMIETOX, aimed at CAVs (Poison Control Centres) and PSPs (Paediatric emergency room).

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 1 month and 16 years who report to the PSPs or contact by telephone the CAVs participating in the study with acute intoxication (defined as contact with a substance that is toxic per se or in such quantities as to cause a harmful effect on the body or administered by a route not intended for that substance)

Exclusion Criteria:

* not acquired informed consent

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: subject between 1 month and 16 years that has reportet to the PSPs or contact by telephone the CAVs participating in the study with acute intoxication
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2033-04-05 (Estimated); Study Completion 2033-08-05 (Estimated)

PRIMARY OUTCOMES:
Determination of Incidence of intoxication in paediatric children | through study completion, an average of 1 year
  Subjects will be stratified by age and type of assumed toxic substance. The incidence of intoxication in paediatric children will be measured taking the total number of new cases of intoxication and divided that by the sum of the person-time of the at-risk population.
Determination of Prevalence of intoxication in paediatric children | through study completion, an average of 1 year
  Subjects will be stratified by age and type of assumed toxic substance. The prevalence of intoxication in this population will be measured calculating the number of people in the sample with the characteristic of interest, divided by the total number of people in the sample.

CONTACTS AND LOCATIONS:
Locations (31):
- Italy (31):
  - Ospedale Santa Maria Annunziata, Bagno a Ripoli, Firenze
  - Ospedale Del Mugello, Borgo San Lorenzo, Firenze
  - Ospedale G B Morgagni, Forlì, Forlì-Cesena
  - Mater Salutis, Legnago, Verona
  - Ospedale Maggiore, Bologna
  - Ospedale Centrale Bolzano, Bolzano
  - Ospedale Brotzu, Cagliari
  - Ospedale San Giuseppe, Empoli
  - Meyer Children's Hospital IRCCS, Florence
  - Ospedale Misericordia, Grosseto
  - Policlinico Messina, Messina
  - Ospedale San Francesco, Nuoro
  - Ao Padova, Padua
  - Nuovo Ospedale Dei Bambini, Parma
  - Policlinico San Matteo, Pavia
  - Policlinico Pescara, Pescara
  - Ospedale Santa Chiara - Cisanello, Pisa
  - Ospedale San Jacopo, Pistoia
  - Ospedale Civile Santa Maria Degli Angel, Pordenone
  - Ospedale Santo Stefano, Prato
  - Ospedale Infermi, Rimini
  - CAV Gemelli, Roma
  - Policlinico Gemelli, Roma
  - Ospedale Regina Margherita, Torino
  - Santa Chiara, Trento
  - Ulss 2 Marca Trevigiana, Treviso
  - Burlo Garofalo, Trieste
  - Clinica Pediatrica Udine, Udine
  - CAV Veneto, Verona
  - Ospedale Della Donna E Del Bambino, Verona
  - Ospedale San Bortolo, Vicenza